CLINICAL TRIAL: NCT03812601
Title: Biatrial Global High-density Electroanatomical Mapping of Atrial Fibrillation - a Prospective Mechanistic Study
Brief Title: Biatrial Global High-density Electroanatomical Mapping of Atrial Fibrillation
Acronym: BiMap-AF
Status: Completed | Type: Observational
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Tim Betts MD MBChB FRCP, Principle Investigator, Oxford University Hospitals NHS Trust
Other Study IDs: 13608
Record Dates: First submitted 2019-01-14; First posted 2019-01-23 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Simultaneous bi-atrial electroanatomic mapping and ablation — Simultaneous bi-atrial electroanatomic mapping during atrial fibrillation and during pacing from 3 different vectors at varying cycle lengths followed by pulmonary vein isolation and AcQMap guided ablation of non-pulmonary vein mechanisms.

SUMMARY:
This study uses two AcQMap imaging and electroanatomical mapping systems (Acutus Medical) to simultaneously visualise and map patterns of wavefront propagation in both the left and right atria during atrial fibrillation in order to identify mechanisms of rhythm propagation and maintenance and the importance of the interaction of the left and right atria. Mapping will also be performed during pacing from different sites and cycle lengths to identify regions of abnormal conduction that may be related to the maintenance of atrial fibrillation.

DETAILED DESCRIPTION:
Patients undergoing first time catheter ablation for atrial fibrillation with undergo simultaneous bi-atrial mapping using two linked AcQMap imaging and mapping systems from Acutus Medical. Mapping will be performed during AF, sinus rhythm and pacing (following cardioversion if required). Pacing will be undertaken from 3 sites in order to create different vectors of conduction and at varying cycle lengths and coupling intervals in order to identify regions of slow and anisotropic conduction. Patients will then undergo pulmonary vein isolation by radiofrequency ablation followed by ablation of non-pulmonary vein targets at the operators discretion (ablation in line with clinical practice and not as part of the study). Regions of focal firing, rotational or slow conduction during AF will be noted and the interaction between each atria described.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial.
* Male or Female, aged 18 years or above.
* Diagnosed with paroxysmal or persistent atrial fibrillation and planned for a catheter ablation procedure.
* In the Investigator's opinion is able and willing to comply with all trial requirements.

Exclusion Criteria:

* Physical or anatomical barriers to the use of two simultaneous mapping catheters
* Previous cardiac surgery
* Previous ablation (catheter or surgical)
* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Participants who have participated in another research trial involving an investigational medicinal product in the past 12 weeks. (Involvement in any other research trial is not a contraindication per se.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing their first catheter ablation procedure for atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Spatiotemporal distribution of non-pulmonary vein focal impulses identified during non-contact mapping of atrial fibrillation | Catheter ablation procedure
  The number and location of focal impulses will be collected over 2 recordings
Spatiotemporal distribution of irregular and rotational activation during 2 recordings of atrial fibrillation | Catheter ablation procedure
  Number of sites of irregular and rotational activation (LA and RA) and their frequency over time during 2 recordings of atrial fibrillation
Frequency of inter-atrial wavefront propagation during AF | Catheter ablation procedure
  Proportion of wavefronts originating in each atria activating from left to right and right to left and site of inter-atrial conduction

SECONDARY OUTCOMES:
Outcome of AcQMap guided catheter ablation of atrial fibrillation | 12 months
  Freedom from recurrent atrial fibrillation on 12 lead ECG or >30seconds on ambulatory monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Timothy R Betts, MB ChB, MD, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No